CLINICAL TRIAL: NCT07372703
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics of a Single Oral Dose of VV913 Capsules in Chinese Healthy Participants
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics of VV913 Capsules in Chinese Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VV913-01
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VV913 (Experimental)
  Interventions: Drug: VV913 1mg group; Drug: VV913 2mg group; Drug: VV913 4mg group; Drug: VV913 8mg group; Drug: VV913 15mg group; Drug: VV913 25mg group; Drug: VV913 40mg group
- Placebo (Placebo Comparator)
  Interventions: Drug: VV913 1mg group; Drug: VV913 2mg group; Drug: VV913 4mg group; Drug: VV913 8mg group; Drug: VV913 15mg group; Drug: VV913 25mg group; Drug: VV913 40mg group

INTERVENTIONS:
Drug: VV913 1mg group — 6 participants will receive VV913 1mg orally; 2 participants will receive placebo orally.
Drug: VV913 2mg group — 6 participants will receive VV913 2mg orally; 2 participants will receive placebo orally.
Drug: VV913 4mg group — 6 participants will receive VV913 4mg orally; 2 participants will receive placebo orally.
Drug: VV913 8mg group — 6 participants will receive VV913 8mg orally; 2 participants will receive placebo orally.
Drug: VV913 15mg group — 6 participants will receive VV913 15mg orally; 2 participants will receive placebo orally.
Drug: VV913 25mg group — 6 participants will receive VV913 25mg orally; 2 participants will receive placebo orally.
Drug: VV913 40mg group — 6 participants will receive VV913 40mg orally; 2 participants will receive placebo orally.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending-dose study to evaluate the safety, tolerability and pharmacokinetics characteristics of VV913 Capsules in healthy adults.

DETAILED DESCRIPTION:
The study is designed to enroll 56 participants. The study , conducted as a double-blind study, comprise 7 dose groups with 8 participants each. Participants will be randomly assigned to receive either the VV913 Capsules or placebo in a ratio of 6:2. Dose groups are designed as 1 mg, 2 mg, 4 mg, 8 mg, 15 mg, 25 mg, and 40 mg. Based on observed tolerability and safety data or obtained pharmacokinetic data, adjustments are allowed at all dose levels in the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 45 years old, males ;
2. Males weight no less than 50 kg, with body mass index of 19 to 26 kg/m^2;
3. Vital signs examination, physical examination, laboratory examination ,electrocardiogram examination chest CT are normal or considered abnormal without clinical significance by the investigator;
4. Participants who are willing to take proper contraceptive methods during the study and within 3 months after the the last administration;
5. Participants who are able to understand and follow the study protocol and instructions; participants who have voluntarily decided to participate in this study, and sign the informed consent form.

Exclusion Criteria:

1. Participants with hypersensitivity to preparation or any of the excipients;
2. Participants with allergic constitution (such as asthma, urticaria, eczematous dermatitis and other allergic diseases), or have a history of drug or food allergy;
3. Participants with central nervous system, cardiovascular system, gastrointestinal, respiratory system, urinary, hematologic, or metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials; Participants with a history of gastrointestinal conditions that may impair drug absorption (e.g., gastrectomy or small intestine resection, atrophic gastritis, gastrointestinal ulcers or perforations/fistulas, gastrointestinal bleeding, or obstruction);
4. Participants with a history of surgery within 3 months before screening, or have not recovered from surgery, or have an expected surgical plan during the trial;
5. Participants with a blood donation or blood loss ≥ 400 mL within 3 months before screening, or a history of blood product use within 3 months before screening;
6. Participating in any clinical trial and taking clinical trial drugs within 90 days before screening;
7. Participants who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products within 14 days before screening;
8. Participants who have received vaccination within 14 days before screening, or planned to receive any vaccine during the trial or within 1 week after the end of the study;
9. Participants with a history of drug abuse within 1 year before screening or positive urine drug screening within 1 year before screening results (morphine, tetrahydrocannabinol, methamphetamine, dimethylene diphenazine , ketamine, and cocaine);
10. Participants who drink more than 14 standard units or at least twice a day per week within one year before screening (one standard unit equals 200 mL of beer with 5% alcohol or 25 mL of spirits with 40% alcohol content or 85 mL of wine with 12% alcohol content);
11. Participants who smoke more than 5 cigarettes a day within one year before screening;
12. Participants who can't quit smoking or drinking during the trial period;
13. Participants who are positive for hepatitis B virus surface antigen, hepatitis C virus antibody, treponema pallidum antibody or human immunodeficiency virus antibody (Anti-HIV）;
14. Having special requirements for food, unable to observe a unified diet or having dysphagia;
15. Participants who cannot avoid consuming drinks containing xanthine (such as coffee and tea) or foods (such as chocolate and animal liver), or fruits or juices (such as grapefruit, pomelo, mango, and dragon fruit) that may affect drug metabolism，from 48 hours before administration until the end of the study;
16. Participants who cannot tolerate blood collection with intravenous indwelling needles or blood fainting;
17. Participants with difficulty in swallowing capsules;
18. Participants whose female partners plan to conceive within 3 months;
19. The investigator believes that there are other unsuitable factors to participate this trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Cmax | 72 hours after administration
  maximum observed plasma concentration
Tmax | 72 hours after administration
  time at which Cmax occurs
t1/2 | 72 hours after administration
  half life of elimination
AUC0-t | 72 hours after administration
  area under the plasma concentration time curve from time zero to the last measurable concentration
AUC0-∞ | 72 hours after administration
  area under the plasma concentration-time curve from time zero to infinity
Kel | 72 hours after administration
  elimination rate constant
Vd/F | 72 hours after administration
  apparent volume of distribution during the terminal phase
MRT | 72 hours after administration
  mean residence time
CL/F | 72 hours after administration
  apparent clearance
AE & SAE | from day1 to day7 after administration
  Adverse event & serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Principal Investigator — The First Affiliated Hospital of Anhui Medical University

IPD SHARING:
Plan to Share IPD: No